CLINICAL TRIAL: NCT07205991
Title: Assisting Digital HEalth REtention (ADHERE Trial): Protocol for a Study Within a Trial (SWAT)
Brief Title: ADHERE Trial: Strategies to Improve Mobile App Adherence
Acronym: ADHERE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuroscience Research Australia (Other)
Responsible Party: Principal Investigator, James McAuley, Principal Investigator, Neuroscience Research Australia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iRECS4383 - SWAT
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain
Keywords: Back Pain; Digital Health; Hypnosis; Pain Education; Chronic Pain
MeSH Terms: conditions — Low Back Pain; Back Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: The study will randomly allocate participants from the intervention group of the NOTUS Trial into one of three parallel arms in a 1:1:1 ratio.
Masking Description: General practitioners and statisticians will be blind to group allocation. Blinding will be maintained for the entire duration of the trial until all data have been collected, and data analysis and interpretation have been completed. The personnel involved in the daily operations of the trial (e.g., research assistants and investigators who will provide possible technical support to participants and trial managers) will be unblinded to group allocation and will not be involved in the analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- App notifications (Active Comparator): Participants will receive the standard app notifications. Reminders are automatically sent at 8pm each day. A user can change the time of their reminder or turn off reminders in the app. The purpose of the app notifications is to increase motivation to complete the app sessions. An example app notification is: Your path to pain management is just a session away. Have you listened today?
  Interventions: Behavioral: App notifications
- Phone calls (Experimental): Participants will receive standard app notifications, and if they do not engage with the intervention for more than three consecutive days , they will be contacted for adherence with up to two phone calls or voice messages, one week apart. The purpose of these calls will be to increase motivation and assess whether participants are experiencing any difficulties using the app or completing the sessions. We expect the calls to last no longer than five minutes. The phone call will include the following communication: Hi [Name], it's [Researcher] from Neuroscience Research Australia calling about the NOTUS back pain trial. I saw that you've done a few sessions on the NOTUS app - great job! We haven't seen you in the Relio app lately, so I wanted to check in and see if everything is working okay or if you need any help with anything. We look forward to seeing you back on the app as you continue retraining your pain system.
  Interventions: Behavioral: Phone calls
- Text messages (Experimental): Participants will receive the standard app notifications, and if they do not engage with the intervention for more than three consecutive days , they will be contacted for adherence with up to two SMS reminders, one week apart. The purpose of these SMS will be to increase motivation and assess whether participants are experiencing any difficulties using the app or completing the sessions. The text messages will include the following: Hey [Name], this is [Researcher] from Neuroscience Research Australia. I saw that you've done a few sessions on the NOTUS app - great job! We haven't seen you in the Relio app lately, so I wanted to check in and see if everything is working okay or if you need any help with anything. We look forward to seeing you back on the app as you continue retraining your pain system.
  Interventions: Behavioral: Text messages

INTERVENTIONS:
Behavioral: Phone calls — Participants will receive standard app notifications and be contacted for adherence via two phone calls, a week apart, if they fail to engage with the intervention for more than three consecutive days. The purpose of these calls will be to assess whether participants are experiencing any difficulties using the app or completing the sessions.
  Arms: Phone calls
Behavioral: Text messages — Participants will receive the standard app notifications and receive a maximum of 2 text messages (SMS) a week apart, if they fail to engage with the intervention for more than three consecutive days.
  Arms: Text messages
Behavioral: App notifications — Participants will receive the standard app notifications .
  Arms: App notifications

SUMMARY:
This study aims to evaluate the effectiveness of two communication interventions, compared to standard app notifications, in increasing adherence to a mobile health app among individuals with chronic low back pain. The main question it aims to answer is:

Do phone calls or text messages increase adherence compared to app notifications in patients receiving a digital health intervention for chronic back pain?

Participants will:

A) Receive pain education and clinical hypnosis via a mobile app for managing chronic LBP; B) Will be contacted up to twice via phone call or text message, or they will only receive standard notifications from the app.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing non-specific chronic low back pain (LBP), defined as pain between the 12th rib and the buttock crease.
* LBP with or without leg pain (in case of leg pain, LBP is worse than leg pain).
* Currently consulting with a general practitioner for their non-specific chronic LBP across Australia.
* Mean pain intensity score on the Numeric Rating Scale ≥ 3/10 in the past week.
* A score of at least moderate on question 8 of the physical functioning component of the SF-36 questionnaire.
* Access to a mobile device with minimal requirements to download the study app (300MB).
* An internet connection to access the mobile app functionalities.
* Able to understand English via reading and audio materials.
* Randomised to experimental group at NOTUS Trial.

Exclusion Criteria:

* Known or suspected specific spinal (e.g., radiculopathy, fracture) or specific non-spinal non- (e.g., tumour, infection) pathology.
* Less than six months post-spinal surgery.
* Scheduled for major surgery during the program or the follow-up period.
* Known or suspected serious psychiatric condition not being treated by a health professional that would impact adherence to the trial activities.
* Known or suspected sight or hearing problems that would limit access to the intervention components (reading and listening using headphones).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2027-05-26 (Estimated); Study Completion 2028-05-26 (Estimated)

PRIMARY OUTCOMES:
Number of sessions completed | Week 8 post-randomisation
  Mean difference of the number of sessions completed over 8 weeks between groups.

SECONDARY OUTCOMES:
Adherence rate (completer vs. non-completer) | Week 8 post-randomisation
  Participants will be classified as "completers" if they have attended at least 24 sessions (new or repeated) during the 8-week treatment period of the host trial. This threshold represents an average of three clinical sessions per week over 8 weeks.
Missing follow-up rate | Week 8 post-randomisation
  Participants will be classified as "follow-up completer" when they completed all primary, secondary and intermediate measures or as "follow-up missing" when they did not complete all primary, secondary and intermediate measures at the 8-week follow-up.
Withdrawal rate | Week 8 post-randomisation
  Participants will be classified as "withdrawal" if they formally withdrew consent, or as "non-withdrawal" if they remained enrolled in the trial at the 8-week follow-up.
Cost-effectiveness | Week 8 post-randomisation
  The mean difference in costs and adherence between groups will be used to calculate the incremental cost-effectiveness ratio (ICER), representing the average additional cost (expressed in Australian dollars - AUD) required to achieve one additional completed session. This outcome reflects the economic efficiency of each engagement strategy (SMS or phone call) compared to others.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuroscience Research Australia, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available to interested researchers only upon reasonable request and once the proposed research project has received separate ethics approval from a Human Research Ethics Committee.
  Request to the data custodian, the Principal Investigator (j.mcauley@neura.edu.au).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available after the publication of the study reports. There is no end date for the availability of study data.

REFERENCES:
- See also: Related Info — https://doi.org/10.1016/j.sciaf.2024.e02436
- See also: Related Info — https://doi.org/10.1186/s13063-024-08004-0
- See also: Related Info — https://doi.org/10.1016/j.jclinepi.2019.04.009
- See also: Related Info — https://doi.org/10.1016/j.jclinepi.2003.08.009
- See also: Related Info — https://doi.org/10.1136/bmj.h5651
- See also: Related Info — https://doi.org/10.1016/j.jphys.2019.08.005
- See also: Related Info — https://doi.org/10.1136/bmj-2021-067742
- See also: Related Info — https://doi.org/10.1007/s10608-014-9606-z
- See also: Related Info — https://doi.org/10.2196/jmir.1923
- See also: Related Info — https://doi.org/10.1371/journal.pone.0088166
- See also: Related Info — https://doi.org/10.2196/43727
- See also: Related Info — https://doi.org/10.1016/j.jad.2017.12.028
- See also: Related Info — https://doi.org/10.2196/30880
- See also: Related Info — https://doi.org/10.2196/43808
- See also: Related Info — https://doi.org/10.1186/s40885-021-00176-0
- See also: Related Info — https://doi.org/10.1016/j.jgo.2022.06.004
- See also: Related Info — https://doi.org/10.1016/j.janxdis.2016.09.012
- See also: Related Info — https://doi.org/10.4085/1062-6050-43.2.215
- See also: Related Info — https://doi.org/10.2196/56897
- See also: Related Info — https://doi.org/10.1007/s10916-024-02135-2
- See also: Related Info — https://doi.org/10.1371/journal.pone.0203127
- See also: Related Info — https://doi.org/10.1016/j.jpain.2010.06.005
- See also: Related Info — https://doi.org/10.1097/ajp.0000000000001289
- See also: Related Info — https://doi.org/10.2196/38261
- See also: Related Info — https://doi.org/10.1016/j.pec.2013.10.027
- See also: Related Info — https://doi.org/10.1016/s0140-6736(05)17709-5
- See also: Related Info — https://doi.org/10.1016/j.jid.2018.06.165
- See also: Related Info — https://doi.org/10.1213/ane.0000000000004410
- See also: Related Info — https://doi.org/10.1016/S0140-6736(02)07816-9
- See also: Related Info — https://doi.org/10.1186/1471-2288-13-92
- See also: Related Info — https://doi.org/10.1186/s13063-018-2535-5
- See also: Related Info — https://doi.org/10.1016/j.apmr.2023.06.002
- See also: Related Info — https://doi.org/10.1016/j.conctc.2020.100572

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Transparency statement + Protocol + SAP (2026-01-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT07205991/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: Protocol + SAP 2025 (2025-09-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT07205991/Prot_SAP_000.pdf